CLINICAL TRIAL: NCT02141737
Title: Effect of Pre-injection of Lidocaine on Myoclonus Induced by Induction With Etomidate in Elderly Patients During General Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140514
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Lidocaine; Saline Solution; Midazolam; Fentanyl; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group C (Placebo Comparator): Induction protocol: patients will be given 2 ml normal saline solution, 1 minutes later, 0.3 mg/kg etomidate is injected within 30 to 60 s, and 90 s after the injection of etomidate, 0.2 mg/kg midazolam, 3 μg/kg fentanyl, 0.6 mg/kg rocuronium are given sequently.
  Interventions: Drug: Etomidate Fat Emulsion Injection; Drug: normal saline; Drug: Midazolam Injection; Drug: Fentanyl Citrate Injection; Drug: Rocuronium Injection
- Group L1 (Experimental): Induction protocol: patients will be given 2 ml diluted lidocaine injection in which 20 mg lidocaine is contained, 1 minutes later, 0.3 mg/kg etomidate is injected within 30 to 60 s, and 90 s after the injection of etomidate, 0.2 mg/kg midazolam, 3 μg/kg fentanyl, 0.6 mg/kg rocuronium are given sequently.
  Interventions: Drug: Lidocaine Hydrochloride Injection; Drug: Etomidate Fat Emulsion Injection; Drug: normal saline; Drug: Midazolam Injection; Drug: Fentanyl Citrate Injection; Drug: Rocuronium Injection
- Group L2 (Experimental): Induction protocol: patients will be given 2 ml diluted lidocaine injection in which 30 mg lidocaine is contained, 1 minutes later, 0.3 mg/kg etomidate is injected within 30 to 60 s, and 90 s after the injection of etomidate, 0.2 mg/kg midazolam, 3 μg/kg fentanyl, 0.6 mg/kg rocuronium are given sequently.
  Interventions: Drug: Lidocaine Hydrochloride Injection; Drug: Etomidate Fat Emulsion Injection; Drug: normal saline; Drug: Midazolam Injection; Drug: Fentanyl Citrate Injection; Drug: Rocuronium Injection
- group L3 (Experimental): Induction protocol: patients will be given 2 ml lidocaine injection in which 40 mg lidocaine is contained, 1 minutes later, 0.3 mg/kg etomidate is injected within 30 to 60 s, and 90 s after the injection of etomidate, 0.2 mg/kg midazolam, 3 μg/kg fentanyl, 0.6 mg/kg rocuronium are given sequently.
  Interventions: Drug: Lidocaine Hydrochloride Injection; Drug: Etomidate Fat Emulsion Injection; Drug: Midazolam Injection; Drug: Fentanyl Citrate Injection; Drug: Rocuronium Injection

INTERVENTIONS:
Drug: Lidocaine Hydrochloride Injection — Lidocaine injection should be give before the injection of etomidate. In groups L1 and L2, 20 mg and 30 mg lidocaine injection will be diluted to 2ml separately.
  Arms: Group L1; Group L2; group L3
Drug: Etomidate Fat Emulsion Injection — 1 minute after the injection of lidocaine, 0.3 mg/kg etomidate will be given in 30 to 60 s.
  Other Names: Fu Er Li
Drug: normal saline — 2 ml normal saline will be given 1 minute before the injection of etomidate in patients in group C, and in group L1 and L2, normal saline is used to dilute lidocaine injection to 2 ml.
  Arms: Group C; Group L1; Group L2
Drug: Midazolam Injection — 0.02 mg/kg midazolam will be given to the patients in all groups 90 s after the injection of etomidate.
  Other Names: Li Yue Xi
Drug: Fentanyl Citrate Injection — 3 μg/kg fentanyl will be given to patients in all groups after the injection of midazolam.
Drug: Rocuronium Injection — 0.6 mg/kg rocuronium will be given to patients in all groups after the injection of fentanyl.

SUMMARY:
To evaluate the effect of pre-injection of lidocaine on myoclonus induced by induction with etomidate during general anesthesia in elderly patients

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged between 60 and 81 years 2. Body mass index: 20 to 30 kg/m2 3. American Society of Anesthesiology (ASA) Physical Status: Ⅰ or Ⅱ 4. Signed informed consent form

Exclusion Criteria:

* 1. Use of sedatives or opioids 2. History of central nervous system diseases, like epilepsy, shaking palsy, or chorea, etc 3. Hyperthyroidism 4. Serious diabetes 5. Hyperkalemia 6. Cardiac surgery 7. Serious ventricular disease or atrioventricular block 8. Liver or renal dysfunction 9. Allergies to amide local anesthetics or fat emulsion

Ages: 60 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
severity of myoclonus induced by | 90 seconds from the beginning of etomidate injection
  myoclonic movements are graded as 0=no myoclonus, 1=mild myoclonus (short movement of a body segment e.g., a finger or a wrist), 2=moderate myoclonus (mild movement of two different muscle groups e.g., face and arm), or 3=severe myoclonus (intense myoclonic movement in two or more muscle groups, fast adduction of a limb)
intensity of injection pain | during the injection of etomidate, expected to be within 1 minutes
  The intensity of pain was graded using a verbal rating scale. 0-None (negative response to questioning)
  1. Mild pain (pain reported only in response to questioning without any behavioral signs)
  2. Moderate pain (pain reported in response to questioning and accompanied by a behavioral sign or pain reported spontaneously without questioning)
  3. Severe pain (strong vocal response or response accompanied by facial grimacing, arm withdrawl or tears)

SECONDARY OUTCOMES:
hemodynamic parameters after injection of etomidate | baseline to 2 minutes after injetion of etomidate
  Heart rate and mean arterial pressure will be recorded before induction, before the injection of etomidate, 1 minute and 2 minutes after injection of etomidate

CONTACTS AND LOCATIONS:
Locations (1):
- TangDu Hospital,FMMU, Xi’an, Shanxi, China